CLINICAL TRIAL: NCT00728741
Title: Functional Neuro-Imaging of Strategy Use During Human Behavior
Brief Title: Brain Activity During Strategic Planning
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080192; 08-N-0192
Record Dates: First submitted 2008-08-05; First posted 2008-08-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-26

CONDITIONS: Healthy Volunteers
Keywords: Neural Networks; Cortical Activation; Strategy; fMRI; Healthy Volunteer; HV

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will locate areas in the brain that help people devise action plans to carry out complex tasks requiring use of strategy. The ability to plan strategically is impaired in patients who have had a stroke affecting the front parts of the brain. This study will use functional magnetic resonance imaging (fMRI) to examine the activity of different areas of the brain during the formulation and execution of plans.

Right-handed healthy volunteers between 18 and 60 years of age may be eligible for this study. Participants come to the NIH Clinical Center four to five times to complete the following procedures:

Visit 1 - Screening

* Medical history
* Physical and neurological examinations

Visit 2 - MRI brain scan (if one has not been done within the past year)

MRI - This test uses a strong magnetic field and radio waves to obtain images of the brain. The scanner is a metal cylinder surrounded by a magnetic field. The subject lies on a table that can slide in and out of the scanner, wearing earplugs to muffle loud noises that occur during the scanning.

Visits 3 to 5 - Task training sessions and two fMRI scans

Functional MRI involves taking MRI scans while the subject performs a task in order to learn about changes in brain regions that are involved in the performance of the task. Subjects are trained in two tasks (see below) and then perform the tasks while in the MRI scanner.

* Task 1: The subject presses computer keys in response to the direction of arrows shown on the computer screen. The keys are pressed according to a given set of rules the subject is taught.
* Task 2: This task is similar to task 1, but the subject is also asked to remember certain previous actions and responses.

DETAILED DESCRIPTION:
OBJECTIVES

Efficient behavior requires the ability to generalize from previous experiences. This can be achieved by behavioral strategies. We use many behavioral strategies; some strategies have strict S-R associations -stop at the RED light-; others are modifiable -balancing skills of a ballerina that becomes very useful during rock climbing- and serve as abstract strategies that enable solving problems.

Strategy use is common in our behavioral repertoire. A strategy can be defined as a set of computations associated with the act of planning and directing overall operations and movements involved in a task. A behavioral strategy that conscious behaving primates spontaneously adopted in order to maximize their rewards have been well characterized in the literature. These are called "Repeat-Stay"/"Change-Shift" strategy, and were shown to be associated with prefrontal neuronal activity during multi-unit intra-cortical recordings, clearly indicating a special role played by the prefrontal cortex in computing strategy use. It is important to understand how the human brain computes and processes strategies. This study aims at understanding the activation patterns, and neuronal connectivity in the human brain when engaged in tasks that require strategies. We hypothesize that application of strategies to solve tasks would show specifically and significantly increase Blood Oxygenation Dependant (BOLD) signal, particularly the fronto-polar cortex (PFp), ventral and orbitofrontal prefrontal cortex (PFV+o) in the human brains.

STUDY POPULATION

The two experiments described in this protocol may recruit up to 61 (6 for the pilot study) adult healthy volunteers.

DESIGN

The study will consist of functional Magnetic Resonance Imaging (fMRI). The fMRI will consist of two separate experiments: (1) the strategy experiment and (2) the memory control experiment. Data will be analyzed separately for each part of the experiment: Responses to tasks will be collected and this data (response times, accuracy rates) will be searched for statistically significant differences using linear contrasts in an ANOVA model.

The imaging fMRI data will be analyzed for statistically significant functional activations by using an implementation of the General Linear Model (GLM) (R. Turner et al., 1998; K. J. Friston et al., 2005) in Statistical Parametric Mapping (SPM).

OUTCOME MEASURES

We propose to acquire response data (response times, error rates), and functional brain activation data using fMRI. Therefore, we would have two outcome measures.

From the response data we will evaluate statistically significant differences in response times, error rates, learning curves.

From the BOLD fMRI data, the main outcome would be task specific neural activations that would regress with the behavioral tasks in a General Linear Model.

These measures will further our understanding about how the human brains use strategies during complex task performance. This will lay the foundation to our understanding for how we are capable of generalizing our experiences from specific instances. Such knowledge will also improve our understanding of various aspects of movement genesis, and is likely to eventually shed light on various movement disorders including psychogenic movement disorders and chorea among others.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects from ages 18 to 60
* Subjects must be right-hand dominant as defined by the Edinburgh Handedness inventory: (R. C. Oldfield, 1971) -Right lateralized handedness quotient of greater than 0.75 will be considered R handed)
* Subjects willing to abstain from caffeine or alcohol for 48 hours prior to the FMRI scanning.

EXCLUSION CRITERIA:

* Subjects with clinically significant abnormal findings on neurological exam in any of the following neurological domains: cognitive, cranial nerve, motor, sensory, cerebellar functions.
* Subjects who are pregnant (as determined by positive urine pregnancy test)
* Subjects with any finding on the MRI safety questionnaire which prevents them from safely undergoing an MRI scan
* Subjects with metallic dental fillings which are likely to cause MRI artifacts
* Subjects with any history of brain tumor, stroke, head trauma or a vascular malformation as obtained by history or from imaging studies
* Subjects with any history of a severe medical condition, such as cardiovascular disease, which would prevent them from lying flat for up to 120 minutes
* Subjects without the capacity to give informed consent
* Subjects with claustrophobia or other restrictions which prevent them from undergoing a scan in a confined space for up to 60 minutes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08-01; Study Completion 2010-05-26

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Blakemore SJ, Goodbody SJ, Wolpert DM. Predicting the consequences of our own actions: the role of sensorimotor context estimation. J Neurosci. 1998 Sep 15;18(18):7511-8. doi: 10.1523/JNEUROSCI.18-18-07511.1998. PMID 9736669
- [Background] Bunge SA. How we use rules to select actions: a review of evidence from cognitive neuroscience. Cogn Affect Behav Neurosci. 2004 Dec;4(4):564-79. doi: 10.3758/cabn.4.4.564. PMID 15849898
- [Background] Bunge SA, Wright SB. Neurodevelopmental changes in working memory and cognitive control. Curr Opin Neurobiol. 2007 Apr;17(2):243-50. doi: 10.1016/j.conb.2007.02.005. Epub 2007 Feb 23. PMID 17321127